CLINICAL TRIAL: NCT02430818
Title: Comparing the Effectiveness of Low-dose Ketamine With Morphine to Treat Pain in Patients With Long Bone Fractures
Brief Title: Comparing Ketamine and Morphine in the Treatment of Acute Fracture Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: were not able to enroll patients to a satisfactory level
Sponsor: Washington University School of Medicine (Other)
Collaborators: MOCEP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201501068
Record Dates: First submitted 2015-04-25; First posted 2015-04-30 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-04

CONDITIONS: Acute Pain; Fractures
Keywords: ketamine; emergency medicine; orthopedics
MeSH Terms: conditions — Acute Pain; Fractures, Bone | interventions — Ketamine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Ketamine is a dissociative agent that is thought to modulate pain by binding to NMDA receptors. Participants assigned to the ketamine arm will be given 0.4 mg/kg IV of ketamine (40 mg maximum).
  Interventions: Drug: ketamine
- Morphine (Experimental): Morphine is an opioid that acts on opioidergic receptors to modulate pain. Participants in the opioid arm will receive 0.1 mg/kg IV of morphine (10 mg maximum).
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: ketamine
  Arms: Ketamine
Drug: morphine
  Arms: Morphine

SUMMARY:
Opioid pain medications such as morphine and dilaudid are commonly used in emergency departments to treat pain in patients. Physicians are familiar with the side effects of these medications; the most concerning of which is slowing or stopping a patient's breathing, as well as dangerously lowering their blood pressure. An alternative medication is ketamine. This medication is also commonly used in the emergency department, although it is typically used to help sedate patients for uncomfortable procedures. Ketamine has also been used for pain control, but in a much lower dosage that does not sedate patients. When used for analgesia, it has typically been administered in combination with opioid pain medications. To date, there is no study that looks at the effectiveness and safety of using a low dose ketamine alone in comparison to the use of morphine. The purpose of this study is to measure how well low-dose ketamine treats pain compared to morphine and to look at how often serious side effects are seen with each medication.

DETAILED DESCRIPTION:
Opioid analgesia is the standard of care for treating moderate to severe pain in the emergency department. It is an effective medication that most practitioners are familiar using. Opioid use is not without risk, however. In managing acute pain, patients may experience hypotension, respiratory depression, hypoxia, nausea and vomiting, dysphoria, and itching. Patients at risk for respiratory depression include those with advanced age, renal failure, or treated with multiple other sedatives.

The current recommended dose for opioid administration for acute pain management is approximately 0.1 mg/kg as a loading dose, although some sources recommend up to 10 mg for patients weighing more than 50 kg. (Ducharme 2011; Yak 2011) A single center study demonstrated that patients received an average of 0.08 mg/kg of morphine, which did not adequately control their pain; no patient received an initial dose of 10 mg.(Bijur 2012) A post-operative pain study demonstrated that patients needed on average 12 mg or a mean weight-based dose of 0.17 mg/kg of morphine to achieve an acceptable level of pain reduction as determined by a 30 mm change on a visual analog scale.(Aubrun 2003) As such even if patients received 1 mg of hydromorphone, their pain would still not be adequately controlled.

Ketamine is a dissociative anesthetic that is a noncompetitive antagonist of N-methyl-D-aspartate (NMDA) receptors. Low dose ketamine (LDK) (0.03-0.05 mg/kg) has analgesic properties by modulating opioid tolerance and hyperalgesia.(Uprety 2013) Currently, ketamine is used in the emergency department for moderate sedations and "awake" intubations. In the pre-hospital setting, it is used in the management of patients with excited delirium and pain control.(Keseg 2014)(Wiel 2014)(Jennings 2013) Benefits include fewer serious adverse effects, especially involving respiratory depression and hypotension which occurs with high-dose or repeat doses of opioids.(Jennings 2013) In addition to not causing hypotension, ketamine can elevate a patient's blood pressure, which may be useful in some circumstances.(Johansson 2009) Emergence delirium is associated with ketamine; this is a rare adverse event and is usually alleviated with benzodiazepines. Additionally, LDK is unlikely to cause the emergence delirium or the dissociation usually associated with larger doses. Another potential complication is laryngospasm. Fortunately, this too is rare and in most cases, patients are easily bagged through the event.

LDK is efficacious in reducing multiple types of pain in a variety of settings. Ketamine infusions can reduce pain from vaso-occlusive pain crises seen in patients with sickle cell anemia.(Uprety 2013)(Neri 2013)(Jennings 2013) In the postoperative setting and intensive care unit, ketamine reduced the amount of morphine required to control pain.(Galinski 2007)(Bell 2006)(Herring 2013) In out-of-hospital trauma patients, ketamine combined with morphine produced superior analgesia to morphine alone. All patients received morphine and were then randomized to receive either morphine or ketamine if further analgesia was required. Ketamine had a change in the visual analog scale (VAS) of -5.6 (CI -6.2 to -5.0) while morphine had had a change of -3.2 (CI -3.7 to -2.7).(Jennings 2012) In another pre-hospital study, ketamine was administered to 1030 patients for pain or anesthesia. No patients incurred ketamine-induced respiratory adverse events.(Bredmose 2009) Preliminary studies have also investigated LDK in the emergency department (ED). Available research mainly consists of retrospective or observational data. In an observational study performed in an urban ED in California, LDK significantly improved patient's pain without adversely effecting blood pressure, heart rate, or respiratory drive. Twenty-four patients over age 18 who received ketamine for any reason were included. Three received ketamine for sedation while the rest received it for analgesia. Most patients received opioids prior to receiving ketamine, although the opioids did not result in improved pain scores. On a scale of 0 to 10, ketamine reduced pain from 8.9 ± 2.1 to 3.9 ± 3.4 (p<0.0001).(Richards 2013) In another observational, ED based study, ketamine used as an analgesic was investigated. Thirty patients with a variety of painful complaints (abdominal pain, back pain, nephrolithiasis, biliary pain, fractures, sickle cell pain) were enrolled. Patients were initially administered a combination of hydromorphone 0.5 mg and ketamine 15 mg with rescue doses of hydromorphone 1 mg available 15 minutes and 30 minutes after the initial dose of analgesia. In 28 patients (93%), there was a clinically significant decrease of 2 or more points on a numerical rating score measured after the initial administration; 14 patients reported pain scores of 0. Fourteen patients refused any additional hydromorphone and 24 patients (80%) either refused additional hydromorphone at 15 minutes or received a dose at 15 minutes but declined a dose at 30 minutes. Dizziness, nausea, headache, and some dissociative effects were reported.(Ahern 2013) Ketamine administered for analgesia in an urban trauma center was retrospectively reviewed in 35 patients. The most common chief complaint was abscess (46%). The median dose of ketamine received was 10 mg (range 5-35 mg); opioids were co-administered in almost all cases (91%). LDK improved pain scores by at least 3 points in 19/35 patients (54%). Eight patients did not receive a post-drug administration pain score.(Lester 2010) A convenience sample of patients was enrolled in an ED based study in British Columbia. Any patients older than 6 years of age presenting with a painful condition were eligible for enrollment. Patients had to have a score of at least 50 on a 100-mm visual analog score (VAS). All patients received 0.5 mg/kg of intranasal (IN) ketamine and could receive a rescue dose of 0.25 mg/kg IN after 10 minutes for VAS > 50. Within 30 minutes, 35 patients (88%) had a decrease in VAS of at least 13 mm. Patient reported satisfaction was a mean of 7 (5-9) on a patient satisfaction scale of 1-10. Dizziness, nausea, and fatigue were all reported.(Andolfatto 2013) IN ketamine was also demonstrated as an effective analgesic in other pediatric and adult ED based studies.(Yeaman 2013)(Yeaman 2014) While ketamine has been studied in the ED, the available research has multiple limitations. Most of it consists of observational or retrospective studies. As such, there could be multiple explanations for their results due to multiple, uncontrolled confounders. In addition, most studies included patients with any painful complaint and did not have a comparison or control group. We plan to conduct a prospective, randomized study of ketamine compared to opioids in long bone fractures.

ELIGIBILITY:
Inclusion Criteria:

* Eligible Long bone fractures. This will include:
* Humerus
* Tibia
* Fibula
* Femur
* Radius
* Ulna

Exclusion Criteria:

* Injuries older than 24 hours
* Avulsion fractures
* History of substance abuse
* History of chronic opioid dependence
* Pregnancy
* Demonstrates signs of intoxication
* Allergic to ketamine or opioids
* Patients unable to consent
* Hemodynamically unstable (SBP >180mmHg or <100mgHg, HR >130bpm, Respiratory rate <10, oxygen saturations <90%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Musisca, MD, Principal Investigator — Physician
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Ahern TL, Herring AA, Stone MB, Frazee BW. Effective analgesia with low-dose ketamine and reduced dose hydromorphone in ED patients with severe pain. Am J Emerg Med. 2013 May;31(5):847-51. doi: 10.1016/j.ajem.2013.02.008. Epub 2013 Apr 18. PMID 23602757
- [Background] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709
- [Background] Aubrun F, Langeron O, Quesnel C, Coriat P, Riou B. Relationships between measurement of pain using visual analog score and morphine requirements during postoperative intravenous morphine titration. Anesthesiology. 2003 Jun;98(6):1415-21. doi: 10.1097/00000542-200306000-00017. PMID 12766651
- [Background] Bell RF, Dahl JB, Moore RA, Kalso E. Perioperative ketamine for acute postoperative pain. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD004603. doi: 10.1002/14651858.CD004603.pub2. PMID 16437490
- [Background] Bijur PE, Esses D, Chang AK, Gallagher EJ. Dosing and titration of intravenous opioid analgesics administered to ED patients in acute severe pain. Am J Emerg Med. 2012 Sep;30(7):1241-4. doi: 10.1016/j.ajem.2011.06.015. Epub 2011 Sep 9. PMID 21908134
- [Background] Bredmose PP, Lockey DJ, Grier G, Watts B, Davies G. Pre-hospital use of ketamine for analgesia and procedural sedation. Emerg Med J. 2009 Jan;26(1):62-4. doi: 10.1136/emj.2007.052753. PMID 19104109
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Herring AA, Ahern T, Stone MB, Frazee BW. Emerging applications of low-dose ketamine for pain management in the ED. Am J Emerg Med. 2013 Feb;31(2):416-9. doi: 10.1016/j.ajem.2012.08.031. Epub 2012 Nov 16. No abstract available. PMID 23159425
- [Background] Jennings CA, Bobb BT, Noreika DM, Coyne PJ. Oral ketamine for sickle cell crisis pain refractory to opioids. J Pain Palliat Care Pharmacother. 2013 Jun;27(2):150-4. doi: 10.3109/15360288.2013.788599. Epub 2013 May 21. PMID 23692261
- [Background] Jennings PA, Cameron P, Bernard S, Walker T, Jolley D, Fitzgerald M, Masci K. Morphine and ketamine is superior to morphine alone for out-of-hospital trauma analgesia: a randomized controlled trial. Ann Emerg Med. 2012 Jun;59(6):497-503. doi: 10.1016/j.annemergmed.2011.11.012. Epub 2012 Jan 13. PMID 22243959
- [Background] Johansson P, Kongstad P, Johansson A. The effect of combined treatment with morphine sulphate and low-dose ketamine in a prehospital setting. Scand J Trauma Resusc Emerg Med. 2009 Nov 27;17:61. doi: 10.1186/1757-7241-17-61. PMID 19943920
- [Background] Keseg D, Cortez E, Rund D, Caterino J. The Use of Prehospital Ketamine for Control of Agitation in a Metropolitan Firefighter-based EMS System. Prehosp Emerg Care. 2015 January-March;19(1):110-115. doi: 10.3109/10903127.2014.942478. Epub 2014 Aug 25. PMID 25153713
- [Background] Lester L, Braude DA, Niles C, Crandall CS. Low-dose ketamine for analgesia in the ED: a retrospective case series. Am J Emerg Med. 2010 Sep;28(7):820-7. doi: 10.1016/j.ajem.2009.07.023. Epub 2010 Apr 2. PMID 20837262
- [Background] Neri CM, Pestieau SR, Darbari DS. Low-dose ketamine as a potential adjuvant therapy for painful vaso-occlusive crises in sickle cell disease. Paediatr Anaesth. 2013 Aug;23(8):684-9. doi: 10.1111/pan.12172. Epub 2013 Apr 9. PMID 23565738
- [Background] Richards JR, Rockford RE. Low-dose ketamine analgesia: patient and physician experience in the ED. Am J Emerg Med. 2013 Feb;31(2):390-4. doi: 10.1016/j.ajem.2012.07.027. Epub 2012 Oct 4. PMID 23041484
- [Background] Uprety D, Baber A, Foy M. Ketamine infusion for sickle cell pain crisis refractory to opioids: a case report and review of literature. Ann Hematol. 2014 May;93(5):769-71. doi: 10.1007/s00277-013-1954-3. Epub 2013 Nov 15. PMID 24232306
- [Background] Wiel E, Zitouni D, Assez N, Sebilleau Q, Lys S, Duval A, Mauriaucourt P, Hubert H. Continuous Infusion of Ketamine for Out-of-hospital Isolated Orthopedic Injuries Secondary to Trauma: A Randomized Controlled Trial. Prehosp Emerg Care. 2015 January-March;19(1):10-16. doi: 10.3109/10903127.2014.923076. Epub 2014 Jun 16. PMID 24932670
- [Background] Yeaman F, Oakley E, Meek R, Graudins A. Sub-dissociative dose intranasal ketamine for limb injury pain in children in the emergency department: a pilot study. Emerg Med Australas. 2013 Apr;25(2):161-7. doi: 10.1111/1742-6723.12059. Epub 2013 Mar 20. PMID 23560967
- [Background] Yeaman F, Meek R, Egerton-Warburton D, Rosengarten P, Graudins A. Sub-dissociative-dose intranasal ketamine for moderate to severe pain in adult emergency department patients. Emerg Med Australas. 2014 Jun;26(3):237-42. doi: 10.1111/1742-6723.12173. Epub 2014 Apr 8. PMID 24712757

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine: Ketamine is a dissociative agent that is thought to modulate pain by binding to NMDA receptors. Participants assigned to the ketamine arm will be given 0.4 mg/kg IV of ketamine (40 mg maximum).
  ketamine
- Morphine: Morphine is an opioid that acts on opioidergic receptors to modulate pain. Participants in the opioid arm will receive 0.1 mg/kg IV of morphine (10 mg maximum).
  morphine
Period: Overall Study
Arm/Group | Ketamine | Morphine
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Morphine | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 37 [19 to 68] | 46 [19 to 77] | 41 [19 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Pain Treatment-VAS (Visual Analog Scale)
Description: Study outcomes involve change in participants' pain as measured by a visual analog scale. The scale is a 10 inch line from 0 to 10 inches with 10 being the most pain and 0 being no pain. There are no units on the scale; it is just a straight line from no pain (0) to the worst pain (10). We assessed at o, 15, and 60 minutes but only scored the VAS at 60 minutes.
Time Frame: At 0 minutes and 60 minutes
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- Ketamine; Morphine: We asked patients if they would use the study medication again for acute pain.
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 6 | 4
score on a scale | 4 (1.3) | 4 (1.8)

2. Secondary Outcome: Number of Participants With an Adverse Effects
Description: We will monitor for adverse effects and record for changes in vital signs including nausea and vomiting, hypotension, respiratory depression, laryngospasm, and emotional and psychological effects (emergence reactions).
Time Frame: 60 minutes
Population: We will include the number of patients with adverse events. Given the very small sample size and small number of events, we are just including total numbers.
Measure: Number; unit: participants
Groups:
- Ketamine; Morphine: Number of participants with Adverse Events
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 6 | 4
participants | 1 | 1

3. Secondary Outcome: Would the Participant Would Consider Using the Drug Given to Them for Pain Relief in the Future
Description: Patients will be assessed to determine whether the participant would consider using the drug given to them for pain relief in the future. It was measured on a likert scale from 1-5 with 1 being did not like and would not use the drug again to 5 being like and would definitely receive the medication again. There are no units. The numbers below are the total number of patients that completed this answer. This was only asked on patients that received medication as if they did not receive medication the answer would not make sense. The median value is the likert value on a scale of 1-5 with the standard deviation.
Time Frame: 60 minutes
Population: We describe all patients that received medication. One patient randomized to morphine did not receive any study medication as her pain improved after being splinted to the extent that she did not have any pain. Two patients were screened and did not meet criteria for inclusion. We used simple, descriptive statistics.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 7 | 5
units on a scale | 4 (1.3) | 4 (1.8)

ADVERSE EVENTS:
Time Frame: Patients will be monitored for 60 minutes for adverse events from the study medication.
Arm/Group | Ketamine | Morphine
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 1/7 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=7) | Morphine (N=6)
emergence reaction (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT02430818/SAP_000.pdf
  • Study Protocol (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT02430818/Prot_001.pdf